CLINICAL TRIAL: NCT01844479
Title: Multi-material, Layer, and Density Insoles for a Patient-specific Approach to Shear and Pressure Reduction in the Treatment and Prevention of Diabetes-related Foot Ulcer
Brief Title: Multi-layer Insoles for a Patient-specific Approach to Shear and Pressure Reduction in Diabetes-related Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, James Wrobel, DPM, MS, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00059211; HUM00059211 (Other: IRBMED)
Record Dates: First submitted 2013-04-12; First posted 2013-05-01 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot
Keywords: diabetic foot ulcer; diabetic foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard innersole (Active Comparator): Per sequence cross over design. Order of testing innersoles was randomized and each testing condition lasted 15 minutes.
  The industry standard diabetic innersole will be used as the active comparator
  Interventions: Other: Standard innersole
- Diabetic Foot Orthotic (Experimental): The Dynamic Foot Orthosis (DFO) is designed with a rolling link mechanism at the distal 3rd to reduce sliding friction at the metatarsal heads in addition to decreasing compressive forces. The relative sliding motion of two compliant surfaces over each other allows some deformation horizontally and lowers frictional resistance. The DFO addresses the friction element by accommodating the normal sliding and rolling motion at the distal 3rd of the foot during gait. Additionally, the DFO has a silicone layer at the metatarsal head and the remainder of the anterior section made of 2 separated orthotic layers that slide over each other. This provides an articulating surface to provide a relative motion between the orthotic segments while transmitting load.
  Interventions: Device: diabetic foot orthotic

INTERVENTIONS:
Device: diabetic foot orthotic — The Dynamic Foot Orthosis (DFO) is designed with a rolling link mechanism at the distal 3rd to reduce sliding friction at the metatarsal heads in addition to decreasing compressive forces. The relative sliding motion of two compliant surfaces over each other allows some deformation horizontally and lowers frictional resistance. The DFO addresses the friction element by accommodating the normal sliding and rolling motion at the distal 3rd of the foot during gait. Additionally, the DFO has a silicone layer at the metatarsal head and the remainder of the anterior section made of 2 separated orthotic layers that slide over each other. This provides an articulating surface to provide a relative motion between the orthotic segments while transmitting load.
  Other Names: shear reducing innersole
  Arms: Diabetic Foot Orthotic
Other: Standard innersole
  Arms: Standard innersole

SUMMARY:
In this pilot study, the first objective is to bench test a novel shear reducing insole and compare it to current standard insoles and shoes. The second objective is to study twenty-seven insensate diabetes patients with pre-ulcerative foot callus to examine for changes in spatial temporal gait including gait initiation, risk of falling, static and dynamic balance, and plantar temperature response to walking and consecutive plantar stress in both footwear conditions.

DETAILED DESCRIPTION:
Device Description: The Dynamic Foot Orthosis (DFO) is designed with a rolling link mechanism at the distal 3rd. It is designed to reduce sliding friction and torque at the metatarsal heads in addition to decreasing compressive forces that is accomplished by the conventional multi-durometer FOs. The relative sliding motion of two compliant surfaces over each other allows some deformation horizontally and lowers frictional resistance. The DFO addresses the friction element by accommodating the normal sliding and rolling motion at the distal 3rd of the foot during gait. Additionally, the DFO has a silicone layer at the metatarsal head and the remainder of the anterior section made of 2 separated orthotic layers that slide over each other. This provides an articulating surface to provide a relative motion between the orthotic segments while transmitting load.

Study Objectives: In this pilot study, the first objective is to bench test a novel shear reducing insole and compare it to current standard insoles and shoes. The second objective is to study twenty-seven insensate diabetes patients with pre-ulcerative foot callus to examine for changes in spatial temporal gait including gait initiation, risk of falling, static and dynamic balance, and plantar temperature response to walking and consecutive plantar stress in both footwear conditions.

Study Design: This is an interventional study. For objective one, changes in compression stiffness and static coefficients of friction will be measured using a force dynamometer in the lab of Professor Albert Shih. A test platform will be built to evaluate the performance of the shear reduction shoe sole design and characteristic of the force, in two directions parallel (shear) and perpendicular to the ground, and the associated deformation under the steady-state and impulse conditions.

For objective two, diabetes patients presenting to the Michigan Orthotics and Prosthetics Center for fabrication and dispensing of diabetic shoes and innersoles will be invited to participate. Twenty-seven insensate diabetes patients with pre-ulcerative foot callus will be enrolled. Patients will wear body worn sensors (LegSys) to measure changes in spatial-temporal gait and static and dynamic balance parameters prior and post usage of the insoles. To reduce the effects of learning from naïve use of novel footwear, the testing sequence between the experimental and standard footwear will be randomized. We will examine increase on foot temperature over 200 steps of continuous walking using the DFO and using standard insoles. We will also examine if the thermal changes are mediated by autonomic neuropathy as measured by sudomotor function. The footwear testing sequence will be randomized and an acclimatization procedure will be followed in an effort to minimize the potential effects of cumulative plantar temperature responses to walking and footwear conditions. We will also examine static balance by measuring center of mass with eyes open and eyes closed condition.

Outcome Measures: For objective one, the primary endpoints will be the compression stiffness and static coefficients of friction. For objective two, plantar foot temperature changes in regions-of-interest in response to walking 200 steps will be measured in each footwear condition and compared to baseline. Other outcome measures include gait analysis, including gait initiation, gait speed, double support time, medial and lateral center of mass displacement, and inter-cycle variability under single and dual task conditions. This will be measured during each footwear condition. Static balance will also be measured in each footwear condition. Using the Romberg's test, we will also assess center of mass displacement and reciprocal hip and ankle motion under eyes open and closed conditions. Sudomotor function will be measured by electrical sweat conductance (ESC), as expressed in microSiemens (µS).

Safety Evaluation: All subjects who sign the informed consent form and are determined to be eligible for treatment will be included in the analysis of safety. Collection, classification and summary analysis of adverse events will be performed.

Duration of Participation: One visit lasting approximately 1 hour.

Duration of Study: One year

Inclusion Criteria: Patients will be included if they have diabetes and have been referred for diabetic shoes. They will also be insensate with pre-ulcerative plantar callus or previous plantar foot ulcer.

Exclusion Criteria: Patients will be excluded if they are unable to independently walk 100 feet, lower extremity prosthesis user, have active cellulitis, foot ulcer, or Charcot foot.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they have diabetes and have been referred for diabetic shoes. They will also be insensate with pre-ulcerative plantar callus or previous plantar foot ulcer.

Exclusion Criteria:

* Patients will be excluded if they are unable to independently walk 100 feet, lower extremity prosthesis user, have active cellulitis, foot ulcer, or Charcot foot.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Wrobel, DPM, MS, Principal Investigator — UMHS
Locations (1):
- Michigan Orthotics and Prosthetics, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Belmont B, Wang Y, Ammanath P, Wrobel JS, Shih A. An apparatus to quantify anteroposterior and mediolateral shear reduction in shoe insoles. J Diabetes Sci Technol. 2013 Mar 1;7(2):410-9. doi: 10.1177/193229681300700218. PMID 23567000
- [Result] Wrobel JS, Ammanath P, Le T, Luring C, Wensman J, Grewal GS, Najafi B, Pop-Busui R. A novel shear reduction insole effect on the thermal response to walking stress, balance, and gait. J Diabetes Sci Technol. 2014 Nov;8(6):1151-6. doi: 10.1177/1932296814546528. Epub 2014 Aug 7. PMID 25107709

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Innersole Followed by DFO: The industry standard diabetic innersole will be used as the active comparator
  Standard innersole
  DFO The Dynamic Foot Orthosis (DFO) is designed with a rolling link mechanism at the distal 3rd to reduce sliding friction at the metatarsal heads in addition to decreasing compressive forces. The relative sliding motion of two compliant surfaces over each other allows some deformation horizontally and lowers frictional resistance. The DFO addresses the friction element by accommodating the normal sliding and rolling motion at the distal 3rd of the foot during gait. Additionally, the DFO has a silicone layer at the metatarsal head and the remainder of the anterior section made of 2 separated orthotic layers that slide over each other. This provides an articulating surface to provide a relative motion between the orthotic segments while transmitting load.
- Diabetic Foot Orthotic Followed by Standard Innersole: The Dynamic Foot Orthosis (DFO) is designed with a rolling link mechanism at the distal 3rd to reduce sliding friction at the metatarsal heads in addition to decreasing compressive forces. The relative sliding motion of two compliant surfaces over each other allows some deformation horizontally and lowers frictional resistance. The DFO addresses the friction element by accommodating the normal sliding and rolling motion at the distal 3rd of the foot during gait. Additionally, the DFO has a silicone layer at the metatarsal head and the remainder of the anterior section made of 2 separated orthotic layers that slide over each other. This provides an articulating surface to provide a relative motion between the orthotic segments while transmitting load.
  The industry standard diabetic innersole will be used as the active comparator
  Standard innersole
Period: First Intervention up to 30 Minutes
Arm/Group | Standard Innersole Followed by DFO | Diabetic Foot Orthotic Followed by Standard Innersole
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Second Intervention up to 30 Minutes
Arm/Group | Standard Innersole Followed by DFO | Diabetic Foot Orthotic Followed by Standard Innersole
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: The industry standard diabetic innersole will be used as the active comparator
  Standard innersole
  The Dynamic Foot Orthosis (DFO) is designed with a rolling link mechanism at the distal 3rd to reduce sliding friction at the metatarsal heads in addition to decreasing compressive forces. The relative sliding motion of two compliant surfaces over each other allows some deformation horizontally and lowers frictional resistance. The DFO addresses the friction element by accommodating the normal sliding and rolling motion at the distal 3rd of the foot during gait. Additionally, the DFO has a silicone layer at the metatarsal head and the remainder of the anterior section made of 2 separated orthotic layers that slide over each other. This provides an articulating surface to provide a relative motion between the orthotic segments while transmitting load.
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Full Range); unit: years] | 65.1 [38 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Plantar Foot Temperature Changes in Regions-of-interest in Response to Walking
Description: Plantar foot temperature changes in regions-of-interest in response to walking 200 steps will be measured in each footwear condition and compared to baseline.
Time Frame: baseline and after 200 steps in each condition, this is a single visit study expected to last one hour
Measure: Mean (Standard Deviation); unit: Absolute change in temperature degrees
Groups:
- Standard Innersole: The industry standard diabetic innersole will be used as the active comparator
  Standard innersole
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
Absolute change in temperature degrees | 0.758 (1.48) | 0.272 (1.21)

2. Secondary Outcome: Gait Initation - Single Task
Description: The number of steps taken to reach steady state walking under single task. Single task means walking without a simultaneous mental task.
Time Frame: during each foot wear condition up to 30 minutes
Measure: Mean (Standard Deviation); unit: Number of steps
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
Number of steps | 4.53 (0.63) | 4.32 (0.58)

3. Other Pre Specified Outcome: Stride Velocity - Single Task
Description: Stride velocity steady state gait single task. Single task means walking without a simultaneous mental task.
Time Frame: during each foot wear condition up to 30 minutes
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
meters/second | 1.08 (0.005) | 1.10 (0.004)

4. Other Pre Specified Outcome: Sudomotor Function
Description: Sudomotor function will be measured by electrical sweat conductance (ESC), as expressed in microSiemens (µS).
Time Frame: at baseline, this is a single visit study expected to last one hour
Measure: Mean (Standard Deviation); unit: µS
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
µS | 70.15 (11.43) | 70.15 (11.43)

5. Secondary Outcome: Gait Initiation - Dual Task
Description: The number of steps taken to reach steady state walking under dual task. Dual task used a simultaneous mental task while walking.
Time Frame: during each foot wear condition up to 30 minutes
Measure: Mean (Standard Deviation); unit: Number of steps
Groups:
- Standard Innersole: Per sequence cross over design. Order of testing innersoles was randomized and each testing condition lasted 15 minutes.
  The industry standard diabetic innersole will be used as the active comparator
  Standard innersole
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
Number of steps | 3.58 (0.53) | 3.42 (0.58)

6. Secondary Outcome: Stride Velocity - Dual Task
Description: Stride velocity during steady state dual task. Dual task used a simultaneous mental task while walking.
Time Frame: during each foot wear condition up to 30 minutes
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
m/s | 1.01 (0.05) | 1.00 (0.04)

7. Secondary Outcome: Double Support Time Single Task
Description: percentage of stride time spent in double support time during gait initiation. Double support time refers to the time spent with both feet on the ground. Single task means walking without a simultaneous mental task.
Time Frame: during each foot where condition up to 30 minutes
Measure: Mean (Standard Deviation); unit: percentage of stride time
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
percentage of stride time | 31.6 (2.4) | 28.3 (1.3)

8. Secondary Outcome: Double Support Time Dual Task Gait Initiation
Description: percentage of stride time spent in double support time during dual task conditions and during gait initiation. Double support time refers to the time spent with both feet on the ground. Dual task used a simultaneous mental task while walking.
Time Frame: during each foot where condition up to 30 minutes
Measure: Mean (Standard Deviation); unit: percentage of stride time
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
percentage of stride time | 31.5 (2.2) | 29.8 (1.3)

9. Secondary Outcome: Medial and Lateral Center of Mass Displacement Single Task
Description: Mediolateral (side-to-side) center of mass displacement with displacement in deg2 (degrees squared) under single task gait conditions. Single task means walking without a simultaneous mental task.
Time Frame: under each foot where condition up to 30 minutes
Measure: Mean (Standard Deviation); unit: deg2
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
deg2 | 4.60 (0.48) | 4.61 (0.36)

10. Secondary Outcome: Medial and Lateral Center of Mass Displacement Dual Task
Description: Mediolateral (side-to-side) center of mass displacement in deg2 (degrees squared) under dual task gait. Dual task used a simultaneous mental task while walking.
Time Frame: both footwear conditions up to 30 minutes
Measure: Mean (Standard Deviation); unit: deg2
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
deg2 | 4.73 (0.65) | 3.99 (0.3)

11. Secondary Outcome: Gait Speed Variability Single Task
Description: Gait speed variability (estimated using coefficient and variation of stride velocity) Single task means walking without a simultaneous mental task.
Time Frame: both footwear conditions up to 30 minutes
Measure: Mean (Standard Deviation); unit: percentage of gait
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
percentage of gait | 6.8 (2.3) | 5.5 (2.1)

12. Secondary Outcome: Gait Speed Variability Dual Task
Description: Gait speed variability (estimated using coefficient and variation of stride velocity) Dual task used a simultaneous mental task while walking.
Time Frame: Both footwear conditions up to thirty minutes
Measure: Mean (Standard Deviation); unit: percentage of gait
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Number analyzed (Participants) | 27 | 27
percentage of gait | 7.45 (2.69) | 5.08 (0.97)

ADVERSE EVENTS:
Arm/Group | Standard Innersole | Diabetic Foot Orthotic
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No